CLINICAL TRIAL: NCT00818103
Title: Characteristic Study on Chinese Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Professor Hu Xueqiang, The Third Affiliated Hospital of Sun Yat-sen University, Department of Neurology
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2007027; 2007027
Expanded Access: Available
Record Dates: First submitted 2008-12-31; First posted 2009-01-07 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis,Genetics,Pathogenesis,Pathology,Therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Atorvastatin

ARMS (1):
- Atorvastatin, β-interferon, EPO (Experimental)
  Interventions: Drug: atorvastatin; Drug: β-interferon; Drug: EPO

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin 40mg p.o. qn for 2 years
Drug: β-interferon — β-interferon 50ug i.m. qod for 2 years
Drug: EPO — EPO 10000U i.h. bid for 5 days

SUMMARY:
Compared with MS in white populations, in people of China descent multiple sclerosis (MS)is characterized by lower prevalence, more frequent and severe involvement of the visual system at onset and during the entire clinical course, more common occurrence of optic and spinal involvement, relatively rapid progression and less common occurrence of a progressive course. Data are not available for mainland China that are focused on characteristic studies of MS. In this study, the investigators sought to explore the characteristics of MS among Chinese in China, by conducting a study on genetics, pathogenesis, pathology, neuroimaging characteristics, and so on. Based on these data, the investigators try to explore the difference in neuromyelitis optical (NMO) and MS and provide clinical data for treatment guidelines for NNO and MS.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for neuromyelitis optical

  * Optic neuritis
  * Acute myelitis
* At least two of three supportive criteria:

  * Contiguous spinal cord MRI lesion extending over >= 3 vertebral segments
  * Brain MRI not meeting diagnostic criteria for multiple sclerosis
  * NMO-IgG seropositive status
* Criteria for multiple sclerosis:

  * Two or more attacks; objective clinical evidence of two or more lesions, OR
  * Two or more attacks; objective clinical evidence of one lesion, dissemination in space, demonstrated by: MRI or two or more MRI-detected lesions consistent with MS plus positive CSF or wait further clinical attack implicating a different site, OR
  * One attack; objective clinical evidence of two or more lesions, dissemination in time, demonstrated by: MRI or second clinical attack, OR
  * One attack; objective clinical evidence of one lesion (monosymptomatic presentation; clinically isolated syndrome), dissemination in space, demonstrated by: MRI or two or more MRI-detected lesions consistent with MS plus positive CSF and dissemination in time, demonstrated by: MRI or second clinical attack, OR
  * Insidious neurological progression suggestive of MS, one year of disease progression (retrospectively or prospectively determined) and two of the following:

    1. Positive brain MRI (nine T2 lesions or four or more T2 lesions with positive VEP)
    2. Positive spinal cord MRI (two focal T2 lesions)
    3. Positive CSF

Exclusion Criteria:

* > 65 yrs old
* Heavy damage of heart, lung, liver, renal function
* Late neuromyelitis optical or EDSS > 6.0
* Serious hypertension and diabetes
* Serious mental disorders and depression
* Allergic to drug: atorvastatin, β-interferon, EPO, immunoglobulin

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The recurrence of NMO or MS | 1 year

SECONDARY OUTCOMES:
EDSS scores, active lesion detected by MRI | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, The Third Affilated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Zhang B, Jiang Y, Yang Y, Peng F, Hu X. Correlation between serum thyroxine and complements in patients with multiple sclerosis and neuromyelitis optica. Neuro Endocrinol Lett. 2008 Apr;29(2):256-60. PMID 18404143
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19300400?ordinalpos=3&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum